CLINICAL TRIAL: NCT01248169
Title: Impedance Cardiographic Assessment of Gravidas With Severe Hypertension (ICASH)to Assess Impact of Standard Therapy on Hemodynamic Parameters - A Pilot Study
Brief Title: Impedance Cardiographic (ICG) Assessment of Pregnant Women With Severe Hypertension to Assess Impact of Standard Therapy
Acronym: ICASH
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, James Martin, Professor, Ob-Gyn, University of Mississippi Medical Center
Other Study IDs: 2007-0187
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Pregnancy; Proteinuria, With Hypertension (Severe Pre-eclampsia); Delivery; Proteinuria, With Gestational Hypertension (Pre-eclampsia, Severe); Pregnancy; Hypertension, Gestational Hypertension, With Albuminuria (Severe Pre-eclampsia)
MeSH Terms: conditions — Proteinuria; Pre-Eclampsia; Hypertension; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — One tube of blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hydralazine: This group will receive administration of the antihypertensive Hydralazine for the attempted control of their blood pressure and stabilization of their hemodynamic state.
- Labetalol: This group will receive administration of the antihypertensive Labetalol for the attempted control of their blood pressure and stabilization of their hemodynamic state.

SUMMARY:
The utilization of external cardiohemodynamic patient assessment, applying non-invasive stick-on contact patches to the mother's neck on either side and chest wall on either side, enables the practitioner to have information about the patient's cardiac function and vascular status beyond simply blood pressure and pulse. This information, once collected, should open the practitioner's eyes to better assess the patient's disease status and her response to therapy. We will use this information to compare the effectiveness of the two standard medications used for treatment of maternal high blood pressure.

DETAILED DESCRIPTION:
Pregnant patients with severe acute hypertension due either to superimposed preeclampsia, severe preeclampsia or severe gestational hypertension will be randomized to receive either of two antihypertensive agents (hydralazine or labetalol). Just before drug administration and immediately thereafter impedance cardiography of the patient will be undertaken and the results analyzed relative to the cardiac profile and the drug administered to reduce the severe hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous or parous patients with severe hypertension
* Singleton gestation
* Gestational age greater than 20 weeks

Exclusion Criteria:

* Multiple gestation
* Gestational age less than 20 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nulliparous or parous patients with severe hypertension, a singleton gestation, gestational age greater than 20 weeks along who are admitted to the Wiser Hospital for Women and Infants at the University of Mississippi Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Usefulness of Impedance Cardiography (ICG) in pregnant women with hypertension | 36
  ICG test is performed on pregnant women before receiving any antihypertensive medication. Labetalol and Hydralazine, two ot the most commonly used antihypertensives to treat high blood pressure in pregnant women will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: James N Martin, MD, Principal Investigator — SOM-Obstetrics & Gynecology
Locations (1):
- Wiser Hospital for Women and Infants at the University of Mississippi Medical Center, Jackson, Mississippi, United States